CLINICAL TRIAL: NCT00816387
Title: Fallopian Tube Sperm Perfusion (FSP) Versus Intra-uterine Insemination (IUI) in Natural Cycle: a Prospective Randomized Study
Brief Title: Fallopian Tube Sperm Perfusion (FSP) Versus Intra-uterine Insemination (IUI) in Natural Cycle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Burlo Garofolo (Other)
Responsible Party: Giuseppe Ricci, IRCCS Burlo Garofolo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RU01/07
Record Dates: First submitted 2008-12-31; First posted 2009-01-01 (Estimated); Last update posted 2010-12-03 (Estimated); Status verified 2009-03

CONDITIONS: Insemination, Artificial

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IUI (Active Comparator): Intrauterine insemination using standard catheter
  Interventions: Procedure: Intrauterine insemination using standard catheter
- FSP (Experimental): Fallopian tube sperm perfusion using a commercial device for hysterosalpingography and tubal hydropertubation
  Interventions: Procedure: Fallopian tube sperm perfusion

INTERVENTIONS:
Procedure: Fallopian tube sperm perfusion — Patients are treated with fallopian tube sperm perfusion
  Other Names: Cervical cup
  Arms: FSP
Procedure: Intrauterine insemination using standard catheter — Patients are treated with standard intrauterine insemination
  Other Names: Balloon catheter
  Arms: IUI

SUMMARY:
The purpose of this study is to evaluate the efficacy of fallopian sperm perfusion (FSP) in comparison with standard intrauterine insemination (IUI) in natural cycle for couples with unexplained infertility or mild male factor.

DETAILED DESCRIPTION:
A number of randomised controlled trials have been published comparing the efficacy of FSP with standard IUI. A recent meta-analysis has suggested that in couples with unexplained infertility Fallopian tube sperm perfusion together with controlled ovarian hyperstimulation (COH) leads to increased pregnancy rates than IUI and COH. No study has been published comparing the two insemination techniques in natural cycle.

ELIGIBILITY:
Inclusion Criteria:

* infertility for at least 2 years
* age <40 years
* unexplained infertility or mild male factor

Exclusion Criteria:

* previous assisted reproduction treatment

Ages: 24 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 400 (Estimated)
Dates: Start 2007-10; Primary Completion 2009-10 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
clinical pregnancy rate | 2 years

SECONDARY OUTCOMES:
Abortion rate | 2 years
Ectopic pregnancy rate | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Ricci, MD, Principal Investigator — IRCCS Burlo Garofolo
Locations (1):
- IRCCS Burlo Garofolo, Trieste, Italy